CLINICAL TRIAL: NCT04020159
Title: Global Registry for COL6-related Dystrophies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18/NE/0243; 8451 (Other: The Newcastle upon Tyne Hospitals NHS FT)
Record Dates: First submitted 2019-06-28; First posted 2019-07-15 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Bethlem Myopathy; Ullrich Congenital Muscular Dystrophy 1, Digenic, Col6A1/Col6A2; Ullrich Congenital Muscular Dystrophy 1, Autosomal Recessive; Ullrich Congenital Muscular Dystrophy 1, Autosomal Dominant; Bethlem Myopathy 1, Autosomal Recessive; UCMD; BTHLM1
MeSH Terms: conditions — Bethlem myopathy; Scleroatonic muscular dystrophy; Multiple Pterygium Syndrome, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with COL6-related dystrophy: Participants who have volunteered to participate will complete various questionnaires relating to their condition.
  Interventions: Other: Patient Registry

INTERVENTIONS:
Other: Patient Registry — No intervention/treatment

SUMMARY:
The Global Registry for COL6-related dystrophies (www.collagen6.org) is a database for individuals who have been diagnosed with Bethlem Myopathy, Ullrich Congenital Muscular Dystrophy (UCMD) or an intermediate form of these diseases. The registry team is based at the John Walton Muscular Dystrophy Research Centre at Newcastle University, UK and is part of the TREAT-NMD alliance global network of registries. The registry has been developed in partnership with a number of leading neuromuscular researchers and is funded by the Collagen VI Alliance.

This patient registry will:

* Help identify patients for relevant clinical trials as they become available
* Encourage further research into Collagen 6-related dystrophies
* Provide researchers with specific patient information to support their research
* Assist doctors and other health professionals by providing them with up-to-date information on managing Collagen 6- related dystrophies, to help them deliver better standards of care for their patients

The investigators welcome the registration of:

✓ All patients, with a diagnosis of a COL6-related dystrophy (Bethlem Myopathy, Ullrich Congenital Muscular Dystrophy or Intermediate form) , which has been confirmed via genetic testing or muscle biopsy.

DETAILED DESCRIPTION:
The Global Registry for COL6-related dystrophies (www.collagen6.org) is an international registry for patients with a COL6-related condition; no experimental intervention is involved. Patients will receive information on the most up to date standards of care relating to their disease and may be invited to participate in relevant clinical trials. Their data will be updated annually and stored indefinitely, or until they request their data to be removed.

The data will be collected via a secure online form and stored on a secure server. Data collected from patients will include demographic information, diagnosis, current condition (wheelchair use and motor ability, respiratory function, contractures and scoliosis), family history and quality of life. Further information collected from patients' doctors will include genetics, age of onset, lung function, medication, muscle strength, contractures and muscle MRI findings.

One of the purposes of the Global Registry for COL6-related dystrophies is to define the patient population and disease course, therefore data is collected longitudinally and participants will be invited to update their records on a yearly basis.

Access to the database is limited to named individuals, approved by the Principal Investigator, Professor Volker Straub, and the database curator. The database is password protected, with different levels of access. All database entries and contacts are traceable through an audit trail. A SOP has been formulated to cover administration, management and communication procedures for the database.

Researchers and Industry may ask specific questions of registry data. These questions may be to support academic research, feasibility studies for clinical trials or recruitment for clinical trials. Any enquiries for data will be examined and approved by the registry steering committee. Data released for approved enquiries would be de-identified aggregate data. In the case of recruitment for clinical trials when the registry principle investigator and/or curator believe that a patient meets a trial's inclusion criterion and might benefit from participation in a trial, the patient will be contacted by the curator with general information about the upcoming trial and will be asked to contact their local trial/study centre for more information if they are interested in participating. The patient's name or any other personal information will not be given to researchers or industry. Clinical trials will need to have appropriate IRB/ethics board and steering committee approval although the registry will not endorse any particular trial.

Registry participation in voluntary and participants may decline to participate or withdraw consent for their data to be stored in the Global Registry for COL6-related dystrophies at any time without prejudice.

The protocol, patient information sheets and consent forms, and relevant supporting information has been reviewed and approved by NHS HRA Research Ethics Committee and Newcastle University ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of a COL6-related dystrophy (Bethlem Myopathy, Ullrich Congenital Muscular Dystrophy (UCMD), or an intermediate form of these conditions.

Exclusion Criteria:

* absence of a diagnosis of COL6-related dystrophy
* Bethlem Myopathy Type 2, Ullrich Congenital Muscular Dystrophy 2 and other COL12-related conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Self-referring individuals with a confirmed diagnosis of a COL6-related dystrophy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Patient questionnaire | 12 months
  Patient reported genetic diagnosis, motor and respiratory function, contractures, pain, unplanned admissions, and quality of life updated annually.
Clinician questionnaire | 12 months
  Clinician reported details of current medical condition (ambulatory status, medications, comorbidities) and medical history (first presenting symptoms, age at diagnosis, diagnosis (genetic, MRI and muscle biopsy findings)), updated annually.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Straub, Principal Investigator — Newcastle University
Locations (1):
- Newcastle University, Newcastle upon Tyne, United Kingdom